CLINICAL TRIAL: NCT05674734
Title: Relational Trauma as an Etiological Factor of Neurotic and/or Personality Disorders Training Acceptance 4FM as a New Form of Therapy for These Disorders
Brief Title: 4FM Acceptance Training as the New Form of cPTSD-focused Treatment Based on Existential Analysis
Acronym: A4FM/AE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A4FM/AE
Record Dates: First submitted 2022-12-16; First posted 2023-01-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Trauma
Keywords: cPTSD; complex trauma treatment; 4 Fundamental Motivations; Existential Analysis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4FM/AT (Experimental): 4FM Acceptance Training, therapeutic intervention in the form of an additional to TAU (Treatment-As-Usual) module - 12 (1,5 hour) group meetings in the form of 4FM Acceptance Training at Day Care Units at Institute of Psychiatry and Neurology (IPiN) Mental Health Centre for Mokotów and IPiN.
  Interventions: Behavioral: 4FM Acceptance Training
- 4FM/TAU (No Intervention): Treatment As Usual - 12 group therapy meetings at Day Care Units at IPIN and IPIN Mental Health Centre for Mokotów.

INTERVENTIONS:
Behavioral: 4FM Acceptance Training — 4FM Acceptance Training, therapeutic intervention in the form of an additional to TAU module - 12 (1,5 hour) group meetings in the form of 4FM Acceptance Training at Day Care Units at IPIN Mental Health Centre for Mokotów and IPiN (1 meeting weekly).
  Arms: 4FM/AT

SUMMARY:
Research project entitled "The experience of relational trauma as an important etiological factor of neurotic and/or personality disorders. The 4FM Acceptance training as a new form of therapy for these disorders" assumes the following goals:

1. validation of the Polish version of the International Trauma Questionnaire (ITQ);
2. assessment of prevalence of relational trauma among adult psychiatric patients hospitalized at the Institute of Psychiatry and Neurology;
3. development a new therapeutic intervention - 4FM Acceptance training - based on the methodology of the Existential Analysis;
4. assessment of the impact of the 4FM Acceptance training among patients with cPTSD.

The original therapeutic intervention - 4FM Acceptance training - will be developed based on the methodological assumptions of the 4 Fundamental Motivations (4FM) in the Existential Analysis methodology, developed by Alfried Längle, student of Viktor Frankl, a representative of the Existential Psychology, together with other important representatives, i.e. Rollo May, Irvin Yalom and in Poland prof. Antoni Kępiński.

DETAILED DESCRIPTION:
Relational trauma, related to early childhood traumatic experiences in relationships with caregivers, usually parents, significantly affects the overall functioning of a person in adulthood. It may also contribute to the occurrence of neurotic disorders and/or personality disorders. The ICD-11 classification introduces a new diagnosis related to the experience of relational trauma, i.e., "complex post-traumatic stress disorder - complex PTSD" (6B41, complex Post Traumatic Stress Disorder, cPTSD). It is a separate nosological unit from PTSD (6B40) (ICD-11, 2022).

Relational trauma therapy should differ from that recommended in PTSD, as it often happens that the "burden of the past" affects the present. Existential psychotherapy may be an effective form of treatment. The Existential Analysis, Alfried Längle's theory of motivation, can be used to treat people who have experienced relational trauma and meet the criteria of cPTSD diagnosis. The project will analyze the impact of a new group therapeutic intervention - 4FM Acceptance Training - on improving existential fulfilment, increasing basic hope, and reducing symptoms of anxiety and depression. 4FM Acceptance Training is the intervention including self-regulatory strategies and trauma-focused interventions.

The obtained results will allow for the assessment of: dissemination of relational trauma, alexithymia, dissociation, somatoform dissociation in the context of the attachment style among people with mental disorders. Thus, they will contribute to the verification of the hypothesis of relational trauma as an important etiological factor of personality disorders and / or neurotic disorders; the usefulness of the 4FM Acceptance group training in the therapy of people with relational trauma and cPTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent provide.
2. Stable mental state allowing for reliable completion of the questionnaires.
3. Native Polish language.
4. Meeting the cPTSD diagnosis based on ITQ - International Trauma Questionnaire), self-report questionnaire, Cloitre et al. (2021), Polish version validated within the project.

Exclusion Criteria:

1. No consent to participate in the research.
2. Coexisting addiction to alcohol or psychoactive substances, documented intellectual disability, dementia or organic changes of the central nervous system.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The International Trauma Questionnaire (ITQ; Cloitre et al., 2018, Polish version (PL) validated within this study as the separate task) | Through study completion, up to 2 years, before start of the intervention
  20-item self-report scale to assess the diagnostic criteria for PTSD and CPTSD according to ICD-11 (WHO, 2018), cPTSD is diagnosed if the criteria for PTSD are met - at least 2 scores of one of two symptoms from the symptom clusters - AND criteria for Disturbances in Self-Organization are met - at least 2 scores of one of two symptoms from the symptom clusters
Trauma Experiences Checklist (TEC, Nijenhuis et al., 2002, PL: Pietkiewicz, Tomalski, 2016). | Through study completion, up to 2 years, before start of the intervention
  29-item self-report questionnaire that measures 29 types of potential trauma, including criterion A events of PTSD, to assess the correlations among a wide range of reported traumatic experiences, including emotional neglect, emotional abuse, somatoform, as well as psychological, manifestations of dissociation according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (APA, 1994), possible trauma area severity scores range from 0 to 12 for emotional neglect, emotional abuse, physical abuse, sexual harassment, and sexual abuse, and from 0 to 24 for bodily threat
Toronto Alexithymia Scale (TAS-20, Taylor et al.,1994, PL: Ścigała et al., 2020) | Through study completion, up to 2 years, before start of the intervention
  20-item self-report scale that measures alexithymia, difficulty in identifying and describing emotions, a score below 51 indicates no alexithymia, a score equal to or greater than 61 indicates the presence of alexithymia, scores between 52 and 60 indicate the presence of alexithymia
Dissociative Experiences Scale, (DES-R PL, Dalenberg, Carlson, 2010, PL: Pietkiewicz et al., (2016) | Through study completion, up to 2 years, before start of the intervention
  28-item self-report scale that measures frequency of dissociation, the total score ranges from 0 to 196 in DES-R PL, the cutoff for dissociative disorders is over 71 points
Somatoform Dissociation Questionnaire (SDQ-20 PL, Nijenhuis et al., (1996), PL: Pietkiewicz et al., 2018) | Through study completion, up to 2 years, before start of the intervention
  20-item self-report scale that evaluates the severity of somatoform dissociation, the total score ranges from 20 to 100, the cut-off point to reach the maximum sensitivity and specificity of the tool for dissociative (conversion) disorders is 29.5
Attachment Style Questionnaire (ASQ, Feeney,1994, PL: Żechowski et al., 2014) | Through study completion, up to 2 years, before start of the intervention
  40-item self-report scale that measures the attachment style based on four-dimensions model by Bartholomew and Horowitz, attachment dimensions: secure, fearful, preoccupied and dismissing, on each dimension separately, respondents give answers on a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree)
Brief Psychiatric Rating Scale (BPRS, Overall, Gorham, 1962) | Before treatment, 1st week of intervention (first session)
  The BPRS assesses the level of 18 symptoms by clinicians or researchers to measure psychiatric symptoms such as anxiety, depression, and psychoses, the rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe)
The Existence Scale (ES, Längle et al., 2003, PL researchers of the Medical University of Warsaw II Psychiatric Clinic under the direction of Kokoszka and Längle) | Before treatment, 1st week of intervention (first session)
  46-item self-report questionnaire to assess existential fulfillment, the possible score ranges from 46 to 276 points, a high score corresponds to a high degree of existential fulfillment
Penn State Worry Questionnaire (PSQW, Meyer et al., 1990, PL Janowski, 2007) | Before treatment, 1st week of intervention (first session)
  16-item self-report questionnaire to measure intensity of worry and anxiety, the possible score rages from 16 to 80, higher score corresponds to a higher intensity of worry and anxiety
Center for Epidemiologic Studies Depression Scale-Revised (CESD-R, Eaton et al., 2004, PL: Koziara, 2016) | Before treatment, 1st week of intervention (first session)
  20-item self-report scale to measure symptoms of depression in nine different groups as defined by the APA Diagnostic and Statistical Manual, fifth edition, a higher score means a higher probability of meeting the criteria for depression
Basic Hope Questionnaire (BHI-12, Trzebiński and Zięba, 2003) | Before treatment, 1st week of intervention (first session)
  16-item self-report questionnaire to measure basic hope understood, according to Erikson's theory, as an individual's conviction about the order and sense of the world and its favor for people, the possible score rages from 12 to 60, higher score corresponds to a higher basic hope

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS, Overall, Gorham, 1962) | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  The BPRS assesses the level of 18 symptoms by clinicians or researchers to measure psychiatric symptoms such as anxiety, depression, and psychoses, the rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe)
The Existence Scale (ES, Längle et al., 2003, PL researchers of the Medical University of Warsaw II Psychiatric Clinic under the direction of Kokoszka and Längle) | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  46-item self-report questionnaire to assess existential fulfillment, the possible score ranges from 46 to 276 points, a high score corresponds to a high degree of existential fulfillment
Penn State Worry Questionnaire (PSQW, Meyer et al., 1990, PL Janowski, 2007) | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  16-item self-report questionnaire to measure intensity of worry and anxiety, the possible score rages from 16 to 80, higher score corresponds to a higher intensity of worry and anxiety
Center for Epidemiologic Studies Depression Scale-Revised (CESD-R, Eaton et al., 2004, PL: Koziara, 2016) | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  20-item self-report scale to measure symptoms of depression in nine different groups as defined by the APA Diagnostic and Statistical Manual, fifth edition, a higher score means a higher probability of meeting the criteria for depression
Basic Hope Questionnaire (BHI-12, Trzebiński and Zięba, 2003) | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  16-item self-report questionnaire to measure basic hope understood, according to Erikson's theory, as an individual's conviction about the order and sense of the world and its favor for people, the possible score rages from 12 to 60, higher score corresponds to a higher basic hope

OTHER OUTCOMES:
Clinical Global Impression - Improvement scale (CGI-I), patient | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  7-point self report rating scale to rate symptom severity, treatment response and the efficacy of treatment from patient's perspective
Clinical Global Impression - Improvement scale (CGI-I), psychotherapist | After treatment, 12th week of intervention (last session), report - through study completion, an average of 2,5 years
  7-point self report rating scale to rate symptom severity, treatment response and the efficacy of treatment from psychotherapist's perspective

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Draczyńska, Principal Investigator — Institute of Psychiatry and Neurology; Marta Anczewska, prof., Study Director — Institute of Psychiatry and Neurology; Agnieszka Nowakowska, PhD, Study Chair — Nowowiejski Hospital